CLINICAL TRIAL: NCT04247022
Title: Evaluation of Cutaneous Acceptability and Genital Mucosa Acceptability of a Health Care Product (Intimate Gel), and Interference of Microbiota and pH Around the Vaginal Introit, With Instrumental Evaluation of the Mucosa Hydratation
Brief Title: Evaluation of Gynecological Acceptability of a Health Care Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herbarium Laboratorio Botanico Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: All-SE-ES-074832
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Atrophic Vaginitis; Vaginal Diseases
MeSH Terms: conditions — Atrophic Vaginitis; Vaginal Diseases

STUDY DESIGN:
Intervention Model Description: Clinical trial, single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- female subjects, 18-59 y, healthy (Experimental): 74 female subjects, 18 to 59 years of age, healthy with complaints of vaginal dryness that will receive the heath care product (intimate gel) for home use, under real conditions of use, for 28 ± 2 days.
  Interventions: Other: Health care product (intimate gel)

INTERVENTIONS:
Other: Health care product (intimate gel) — heath care product (intimate gel) for home use, under real conditions of use, for 28 ± 2 days

SUMMARY:
The research will be conducted with a product for use in the intimate region in up to 75 research participants who will use the investigational product for 28 ± 2 days. Will be evaluated and followed up throughout the study by a gynecologist to verify the safety and effectiveness of the product and possible adverse events.

The study will evaluate the non-interference of a topical use product on the intimate area, helping to preserve the natural defenses. In addition, the epithelial hydration and pH of the intimate area will be evaluated.

DETAILED DESCRIPTION:
74 female participants, 18 to 59 years of age, healthy with complaints of vaginal dryness. The subjects will be submitted to gynecological evaluation in which pH measurements, hydration measurements and bacterioscopic collection will be performed. Then they will be guided to answer the questionnaires of Perceived Efficacy and Quality of Sexual Life. Next, participants will receive the product for home use, under real conditions of use, for 28 ± 2 days. After 28 ± 2 days of use, subjects will return to the institute, and undergo further evaluations with the gynecologist. New pH measurements, hydration measurements (chronometry), bacterioscopic collection will be performed and the participants will answer the Perceived Efficacy and Quality of Sexual Life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Health volunteers
* Non-injured mucosa in the test region;
* Agreement to comply with safety guidelines to minimize the risk of contamination to COVID-19;
* Agreement to perform molecular testing to detect COVID-19 to enter the study;
* Agreement to adhere to study procedures and requirements and attend the institute on the day(s) and time(s) determined for the evaluations;
* Ability to consent to their participation in the study;
* Age from 18 to 59 years old (25 participants from 18 to 39 years old, 25 participants from 40 to premenopause and 25 participants in climacteria);
* Female participants;
* Vaginal dryness (slight minimum) - according to questions from the gynecologist.

Exclusion Criteria:

* Participants who belong to the risk group for COVID-19, that is, aged over 60 years, with diabetes, with chronic cardiovascular, renal and respiratory problems, immunosuppressed or other conditions that the physician deems to belong to the risk group;
* Participants who have COVID-19, or who have symptoms indicative of the disease in the last 14 days, such as temperature above 36.8°C, fever, cough, shortness of breath, loss of smell, loss of taste and fatigue;
* Pregnancy or breastfeeding;
* Skin pathology in the area of application of the product;
* Diabetes Mellitus type 1; insulin-dependent diabetes; presence of complications due to diabetes (retinopathy, nephropathy, neuropathy); presence of diabetes-related dermatoses (plantar ulcer, lipoid necrobiosis, annular granuloma, opportunistic infections); history of episodes of hypoglycemia, diabetic ketoacidosis and/or hyperosmolar coma;
* Current use of the following medications for topical or systemic use: corticosteroids, immunosuppressants and antihistamines;
* Skin diseases: vitiligo, psoriasis, lupus, atopic dermatitis;
* History of reaction to the category of the tested product;
* Other diseases or medications that may directly interfere with the study or endanger the health of the research participant.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Perceived Hydration | 28 ± 2 days
  Evaluate the perceived hydration through a subjective questionnaire
Hydration (device) | 28 ± 2 days
  Evaluate the hydration, through a hydration measurements by chronometry.

SECONDARY OUTCOMES:
Natural defenses preservation (pH) | 28 ± 2 days
  pH measurements
Natural defenses preservation (microbiota) | 28 ± 2 days
  bacterioscopic collection

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa Pesquisa Dermato-Cosmética Ltda, Campinas, São Paulo, Brazil